CLINICAL TRIAL: NCT07195760
Title: Delayed IntraCranial Hemorrhage in Oral AntiCoagulant Treated Patients With Mild Traumatic Brain Injury (the dICH-OAC Study)
Brief Title: Delayed IntraCranial Hemorrhage in Oral AntiCoagulant Treated Patients With Mild Traumatic Brain Injury
Acronym: dICH-OAC
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Hanne Christensen, Professor, Consultant Neurologist, Bispebjerg Hospital
Other Study IDs: J-23036221; 2211770 (Other: Danish National Center for Ethics)
Record Dates: First submitted 2023-08-29; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Head Trauma; Head Injury; Delirium; Thrombosis
Keywords: Oral anticoagulants; NOAC; DOAC; Vitamin K antagonist
MeSH Terms: conditions — Craniocerebral Trauma; Delirium; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral anticoagulated: Patients admitted with mild head traume and oral anticoagulation treatment, having a CT performed.
- Platelet inhibited: Patients admitted with mild head traume and antiplatelet treatment, having a CT performed.
- Not on antithrombotics: Patients admitted with mild head trauma, not treated with antithrombotics, having a S100B performed.

SUMMARY:
As a low quality, weak recommendation, it is part of the Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults, that patient with a GCS of 14-15 and anticoagulation therapy and a normal CT should be admitted for observation for at least 24 hours. No data are available on the adverse events related to the observational 24-hour admission. The aim was to evaluate the risk of post-CT hemorrhage as well as the risk of complications to an admission (e.g. deleria, thrombosis due to pause of antithrombotic medications.

DETAILED DESCRIPTION:
As a low quality, weak recommendation, it is part of the Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults, that patient with a GCS of 14-15 and anticoagulation therapy and a normal CT should be admitted for observation for at least 24 hours. No data are available on the adverse events related to the observational 24-hour admission.

Because of this, the investigators aim to evaluate the following outcomes in a cohort of consecutive patients aged 65 or above, admitted at the acute neurological department or emergency room of Bispebjerg Hospital in the Capital Region of Denmark from June 1st 2020 - May 31st 2022 following a mild or minimal head trauma with no intracranial hemorrhage on initial head CT and compare outcomes of patients pre-treated with oral anticoagulants to patients treated with platelet inhibitors and patients without antithrombotic treatment:

* Delayed intracranial hemorrhage within 24 hours and 4 weeks (incl. readmissions)
* Delayed diagnosis of intracranial hemorrhage
* Thrombotic events within 1 week of trauma
* Deliria during admission
* Other injuries with a competing need for admissions at other departments

The overall goal is to add to the evidence in the area, so that there can be sufficient evidence, to potentially update the recommendations in the Scandinavian Guideline for initial management of minimal, mild, and moderate head injuries in adults. This with the hope that the results will benefit not only the health care economy, but also the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Minimal (defined according to the Head Injury Severity Score (HISS (Stein and Spettell 1995)) as GCS 15 without any risk-factors) or Mild head trauma (defined according to the HISS as a GCS score of 14 or 15 with risk factors (e.g. OAC-treatment, GCS = 14, repeated vomiting, loss of consciousness, age ≥ 65 and antiplatelet medication))
* No bleeding on initial head CT description

Exclusion Criteria:

* Other reasons for observation despite normal CT, based on the Scandinavian guidelines for initial management of minimal, mild and moderate head injuries in adults:

  * GCS < 14
  * Post traumatic seizures
  * Focal neurological deficits
  * Clinical sign of depressed or basal skull fracture
  * Shunt-treated hydrocephalus

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The identification of patients for screening will follow the Scandinavian guideline algorithm. The first and second group will be patients in whom the procedure code for computer tomography (CT) of the cerebrum has been recorded and who had a prescription of either a platelet inhibitor or an oral anticoagulant (OAC) on admission. The prescription is transferred from the shared medicines cart to the local system by the admitting physician, with the only exception being if the prescription is immediately suspended on admission, which should only be the case if the patient already stopped taking the medication. The third group will be all the patients in whom a s100b test was performed.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Delayed Intracranial hemorrhage within 24 hours | 24 hours
  Hemorrhage found after initial CT scan but within 24 hours of trauma
Delayed Intracranial hemorrhage within 4 weeks | 4 weeks
  Hemorrhage found after initial CT scan but within 4 weeks of trauma
Thrombotic events | 1 week
  Arterial or venous thrombotic events experienced within one week of trauma
Deliria | During admission = up to 1 week after admission
  Description of deliria during admission for initial head trauma
Other injuries with a competing need for admission at another department | admission = up to 1 week after admission

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, MD, PhD, DMSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg and Frederiksberg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No
Aggregated, summary data are to be shared. However, individual participant data will only be made available as according to local law.